CLINICAL TRIAL: NCT03822988
Title: ACCEPTABILITY AND WRITING FREQUENCY OF ADVANCED DIRECTIVES IN ONCO-DERMATOLOGY PATIENTS
Acronym: PADAONCODERM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS-2018/PADAONCODERM
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Advance Directives; Oncology; Skin Cancer; Melanoma; Skin Lymphoma; Skin Squamous Cell Carcinoma; Metastatic Basal Cell Carcinoma
Keywords: advance directives; Advance care planning; Patient's informed; treatment preferences; skin cancer; dermatology
MeSH Terms: conditions — Neoplasms; Skin Neoplasms; Melanoma; Lymphoma, T-Cell, Cutaneous; Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients accepting to answer to the survey: patients with a skin lymphoma OR melanoma OR advanced skin squamous cell carcinoma OR advanced basal cell carcinoma accepting to answer to the anonymous survey
  Interventions: Other: no intervention, only complete a survey

INTERVENTIONS:
Other: no intervention, only complete a survey — we will ask patients to answer to a survey

SUMMARY:
The law about advance directives is evolving but, in France, few people write it.

Te main endpoint of this research is to estimate the proportion of patients who have written their advance directives or considering doing so in onco-dermatologic population. If this rate remains low, some insights on the reasons will be able to be advanced looking at the point of view and opinion of patients about this topic.

Seconds endpoints are :

For patients against or not planning to write it, understand their reasons

Estimate the proportion of patients requesting information and understand how they would like to receive it.

Investigate a possible association between the stage of the oncological disease and the positioning of the patient concerning advance directives.

ELIGIBILITY:
Inclusion Criteria:

> 18 ya

With one of the diagnoses below:

* Melanoma
* Skin lymphoma
* Meckel Carcinoma
* localy advanced or metastatic Basal cell carcinoma or squamous cell carcinoma

Exclusion Criteria:

Patients not in possession of all of its cognitive abilities Patients who can't read patients who don't speak french

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cf beyond
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-06-20 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Writing by the patient of its advance directives | when the patient complete the survey
  Writing by the patient of his advance directves and, if not writing, positioning of the patient (rather favorable or rather unfavorable) as to the writing of his advance directives.

SECONDARY OUTCOMES:
reason for not writing advance directives | when the patient complete the survey
  In patients who have not written their advance directives: reason for not writing the advance directives.
Patient wishing to be more informed about the adavance directives during its management and, if so, by what means. | when the patient complete the survey

CONTACTS AND LOCATIONS:
Overall Officials: anne-claire bursztejn, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy-Brabois hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No